CLINICAL TRIAL: NCT01147367
Title: Physical Activity Benefits After Breast Cancer: Exploring Cytokine Mechanisms
Brief Title: Physical Activity, Fatigue, Sleep, and Inflammation
Acronym: ABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ROG-SCCI-10-004-1; R21CA135017-01A2 (NIH)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: exercise; breast cancer; physical activity; fatigue; sleep dysfunction; cytokines; muscle strength; inflammation
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue; Parasomnias; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): no physical activity intervention
- Exercise intervention (Experimental): 3 month physical activity intervention involving moderate intensity walking and strength training with resistance bands
  Interventions: Behavioral: 3 month physical activity intervention

INTERVENTIONS:
Behavioral: 3 month physical activity intervention — 3 month physical activity intervention involving moderate intensity walking and strength training with resistance bands
  Other Names: exercise
  Arms: Exercise intervention

SUMMARY:
The purpose of the study is to examine the benefits of physical activity for breast cancer survivors related to muscle strength, tiredness, and sleep quality. Also, the study will determine the potential role of inflammation in these benefits.

DETAILED DESCRIPTION:
Our previous research has shown that increases in physical activity can improve the health and well-being of breast cancer survivors. The current study will determine whether the physical activity increases are adequate for improved health by measuring physical activity (accelerometer and self-report), muscle strength, fatigue, and sleep. Moreover, few studies have examined cytokine changes in cancer survivors after participation in a physical activity behavior change intervention with a mechanistic focus on cytokines which may influence the muscle strength, fatigue, and sleep response to the intervention.

Seventy-four female, breast cancer survivors are being recruited within a 50-miles radius of Springfield, IL. Participants will be in the study for approximately 5 months. Participants will be asked to complete a questionnaire at the beginning of the study and 3 months later. A blood sample will be drawn to determine serum cytokine levels.

Volunteers will be randomly assigned to 1 of 2 study groups. The intervention group will participate in a 3 month physical activity intervention involving moderate intensity walking and strength training with resistance bands.

This randomized controlled trial includes the following study aims:

Study aim 1: The intervention group will be compared with the control group to examine the change in physical activity, muscle strength, fatigue, and sleep dysfunction before and after participation in a physical activity intervention.

Study aim 2: To investigate mechanisms that may underlie the effects of the physical activity intervention on muscle strength, fatigue, and sleep, we will compare the intervention group with the control group in terms of changes in cytokine markers of inflammation and evaluate whether such changes are consistent with and may mediate changes in muscle strength, fatigue, and sleep dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Female, 30 to 70 years of age, with first diagnosis of ductal carcinoma in situ (DCIS) or Stage I or Stage II breast cancer
* If chemotherapy or radiation therapy was received, the patient must be at least 4 weeks status post final primary treatment administration to allow treatment related cytokine changes to resolve. The participant may be taking longer term therapies such as aromatase inhibitors, estrogen receptor modulators, etc.
* If the patient has undergone a surgical procedure, she must be at least 8 weeks post-procedure.
* English speaking
* Medical clearance for participation provided by primary care physician or oncologist
* Postmenopausal
* Average fatigue over the past week of ≥ 3 on a 1 to 10 Likert scale or sleep dysfunction ≥ 1 on a 0 to 3 Likert scale
* Participating, on average, in no more than 20 minutes of physical activity on two or fewer days per week during the past six months
* Willing to abstain from "as needed" medications for 7 days prior to each blood draw. "As needed" medications are defined as any medicine (prescription or over-the-counter) that is taken sporadically as needed for specific complaints rather than taken at regularly scheduled intervals (e.g., daily).

Exclusion Criteria:

* Metastatic or recurrent breast cancer
* Inability to ambulate without assistance
* Unstable angina
* New York Heart Association class II, III, or IV congestive heart failure
* Uncontrolled asthma
* Interstitial lung disease
* Current use of steroids
* Having been told by a physician to only do exercise prescribed by a physician
* Dementia or organic brain syndrome
* Schizophrenia or active psychosis
* Connective tissue or rheumatologic disease [i.e., Systemic lupus erythematosus, rheumatoid arthritis, amyloidosis, Reiter's syndrome, psoriatic arthritis, mixed connective tissue disease, Sjögren's syndrome, progressive systemic sclerosis, CREST syndrome, polymyositis, dermatomyositis, vasculitis, polymyalgia rheumatic, temporal arteritis]
* Anticipates undergoing elective surgery during the duration of the intervention which would interfere with intervention participation (e.g., breast reconstructive surgery).
* Do not live or work less than 50 miles from the study site
* Lack of transportation to the study site
* Changes in usual medications expected during the study time period
* Plan to move residence out of the local area during the 5 months of the study
* Plan to travel out of the local area for vacation during the first 4 weeks of the intervention or plan to travel out of the local area for more than a week during the last 8 weeks of the intervention
* Contraindication to participation in physical activity (i.e., moderate intensity walking and strength training with resistance bands)

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
physical activity | baseline and 3 months
  The intervention group will be compared with the control group to examine the change in physical activity, before and after participation in a physical activity intervention. Participants are in the study for approximately 5 months. Assessments will be conducted at baseline, and following the 3 month exercise intervention.
muscle strength | baseline and 3 months
  The intervention group will be compared with the control group to examine the change in muscle strength before and after participation in a physical activity intervention.
fatigue | baseline and 3 months
  The intervention group will be compared with the control group to examine the change in fatigue before and after participation in a physical activity intervention.
sleep dysfunction | baseline and 3 months
  The intervention group will be compared with the control group to examine the change in sleep dysfunction before and after participation in a physical activity intervention.

SECONDARY OUTCOMES:
inflammatory markers (serum cytokine levels) | baseline and 3 months
  The study will also examine whether changes in inflammatory markers mediate improvements in the outcome measures of muscle strength, fatigue, and sleep dysfunction. Blood samples with no potential for extraction of DNA will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q Rogers, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Result] Rogers LQ, Vicari S, Trammell R, Hopkins-Price P, Fogleman A, Spenner A, Rao K, Courneya KS, Hoelzer KS, Robbs R, Verhulst S. Biobehavioral factors mediate exercise effects on fatigue in breast cancer survivors. Med Sci Sports Exerc. 2014 Jun;46(6):1077-88. doi: 10.1249/MSS.0000000000000210. PMID 24212124
- [Result] Rogers LQ, Fogleman A, Trammell R, Hopkins-Price P, Spenner A, Vicari S, Rao K, Courneya KS, Hoelzer K, Robbs R, Verhulst S. Inflammation and psychosocial factors mediate exercise effects on sleep quality in breast cancer survivors: pilot randomized controlled trial. Psychooncology. 2015 Mar;24(3):302-10. doi: 10.1002/pon.3594. Epub 2014 Jun 11. PMID 24916951